CLINICAL TRIAL: NCT02638870
Title: Colonoscopy-related Pain Predicts the Treatment Response of Amitriptyline in Patients With Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Poong-Lyul Rhee, Prof., Samsung Medical Center
Other Study IDs: 2015-08-109
Record Dates: First submitted 2015-12-20; First posted 2015-12-23 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Amitriptyline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Amitriptyline — This was a prospective, observational study conducted at Samsung Medical Center, Seoul, Korea. Enrolled IBS patients underwent colonoscopy and colonoscopy-related pain score was evaluated. After colonoscopy, all patients received 5 mg amitriptyline once daily at bedtime for the first week and 10 mg for the subsequent 3 weeks. After the intervention period of 4 weeks, the treatment response was determined.

SUMMARY:
Irritable bowel syndrome (IBS) is a functional bowel disorder with recurrent abdominal pain and disordered defecation and is one of the most common gastrointestinal problems. In practice, IBS was frequently diagnosed as an exclusion diagnosis for patients with recurrent abdominal pain without an organic cause. Visceral hypersensitivity is the major contributing factor of abdominal pain in IBS. Accordingly, tricyclic antidepressants (TCAs) are widely used for IBS, especially if abdominal pain is a prominent symptom. Indeed, meta-analysis also exhibits the clinically significant efficacy of low dose TCAs in IBS. Nevertheless, over 40% of IBS patients receiving TCAs had no improvement in symptoms after treatment. Theoretically, if TCAs are used for IBS patients with hypersensitivity, its efficacy could be increased.

Although rectal distension test might be used to identify hypersensitive patients with IBS, it has been used only for clinical research because it is painful for the patient. On the contrary, colonoscopy is frequently performed in IBS patients to rule out organic disease and for the purpose of colorectal cancer screening. In a study by Kim and colleagues, IBS patients reported higher pain score after colonoscopy than non-IBS patients. This has prompted the hypothesis that pain scoring during/after colonoscopy could also segregate IBS patients with visceral hypersensitivity showing better treatment response of TCA than those without.

The aims of the present study were to evaluate the colonoscopy-related pain perception and the treatment response of amitriptyline in IBS patients and to investigate the predictive values of the colonoscopy-related pain scale in identifying IBS patients with a response to amitriptyline treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS according to the Rome III criteria

Exclusion Criteria:

* Inflammatory bowel disease or malignancy on colonoscopy.
* Previous abdominal surgery other than appendectomy or cesarean delivery,
* Major psychiatric disorders or Beck Depression Inventory-II score of ≥19
* Significant cardiopulmonary diseases or any malignancies
* Taking pain modulators including selective serotonin reuptake inhibitors (SSRI) or tricyclic antidepressants
* Polypectomy during colonoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBS according to the Rome III criteria were recruited in the outpatient clinic at Samsung Medical Center. Inclusion criteria were age 18-75 years and no evidence of inflammatory bowel disease or malignancy on colonoscopy.
Sampling Method: Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
treatment response of abdominal pain/discomfort | After the intervention period of 4 weeks, the treatment response was determined.
  The primary outcome was the treatment response of abdominal pain/discomfort. The investigators defined a response when a patient experienced a fall of 30% in abdominal symptom compared to baseline.

SECONDARY OUTCOMES:
treatment responses of urgency of defecation | After the intervention period of 4 weeks, the treatment response was determined.
  The secondary outcomes were the treatment responses of urgency of defecation, bloating, and overall IBS symptoms scores.
treatment responses of bloating | After the intervention period of 4 weeks, the treatment response was determined.
treatment responses of overall IBS symptoms scores | After the intervention period of 4 weeks, the treatment response was determined.

CONTACTS AND LOCATIONS:
Overall Officials: Poong-Lyul Rhee, M.D.,Ph.D., Principal Investigator — Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea